CLINICAL TRIAL: NCT06555718
Title: Examining the Effect of the Peer Support Program Applied to Chronic Kidney Patients on Care Outcomes
Brief Title: Peer Support Program in Chronic Kidney Patient
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATADEK2023-21/765
Record Dates: First submitted 2024-07-30; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Peer Review; Hemodialysis Complication; Nurse's Role; Health-Related Behavior
Keywords: Peer sport; nursing; hemodialysis
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: The study will start after obtaining official institutional permissions. The researcher will examine the profile of patients receiving treatment at the dialysis center. After this stage, the following steps will be followed
Who Masked: Participant
Masking Description: Intervation group (Peer support) Control group (Standart care)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Peer support) (Other): "Peer mentors" will be determined among the participant patients in accordance with the peer mentor guide selection criteria.
  The determined peer mentors will participate in the "Peer Mentor Training Programme".
  Implementation of the research; Peer support programme for the intervention group will be carried out for 10 weeks in accordance with the peer guide-client implementation plan Standard follow-up and training programme will be applied to the control group in accordance with the procedures of the institution.
  The data collection forms used in the research process will be collected at the stages specified in the study flow plan and data entry will be made by the researcher.
  Interventions: Behavioral: The Peer Support Program
- Control group (Standart care) (Other): No intervention will be made by the researcher to the control group. The standard care of the institution will be applied to the patients.
  Interventions: Behavioral: Standart care

INTERVENTIONS:
Behavioral: The Peer Support Program — Implementation of the research; Peer support programme for the intervention group will be carried out for 10 weeks in accordance with the peer guide-client implementation plan. Standard follow-up and training programme will be applied to the control group in accordance with the procedures of the institution.
  Arms: Intervention group (Peer support)
Behavioral: Standart care — The standard care provided by the institution will continue.
  Arms: Control group (Standart care)

SUMMARY:
The main advantage of patient-to-patient peer counseling is that it benefits both the client and the peer mentors as real and authentic experiences are shared. Since both individuals go through similar experiences, they can share common feelings. Although there are studies in the literature showing the effectiveness of peer support groups in different patient groups, studies on chronic kidney disease patients are limited. There are no studies on the effects of these programs on caregivers. This study will be conducted to examine the effects of peer support program applied to chronic kidney patients on patient outcomes and caregivers.

DETAILED DESCRIPTION:
This study was planned to be conducted with a randomized controlled experimental design to examine the effect of the peer support program applied to Chronic Kidney patients on patient outcomes and caregivers.

Patients diagnosed with Chronic Kidney Disease and receiving haemodialysis (HD) as a renal replacement method constitute the population of the study. In the a priori power analysis performed to calculate the number of subjects, the effect size was taken as 1.3 (d) based on reference studies. Accordingly, it was found that 34 subjects should be included in the calculation for the independent two-sample t-test according to 0.95 power and 0.05 alpha. The sample of the study will consist of 25 intervention and 25 control CKDs who fulfil the inclusion criteria, taking into account the dropout status.

ELIGIBILITY:
Inclusion and Exclusion Criteria For Peer Mentor Inclusion Criteria;

* Speaking Turkish
* To be literate
* CKD receiving haemodialysis
* Volunteering
* 18 years of age or older
* Being open to communication and co-operation
* Not having any psychiatric disorder

For Patient Inclusion Criteria;

* Speaking Turkish
* To be literate
* CKD receiving haemodialysis
* Volunteering
* 18 years of age or older
* Not having any psychiatric disorder

Exclusion criteria for all participants

* Being under 18 years of age
* Speaking a language other than Turkish
* Not being able to use a telephone

Losses to follow-up

* Experiencing incompatibility with the second peer mentor or client with whom they are paired for peer mentor and peer client
* Death during the period of intervention or follow-up
* Withdrawal of patient consent
* Clinical problems or difficulties attending appointments that hinder follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Adaptation to the disease. | The scale will be completed before the intervention and at 3, 7 and 9 weeks.
  "End Stage Renal Disease Adaptation Questionnaire (ESRD-AQ)" Total score varies between 0 and 1200. As the score obtained from the scale increases, the level of treatment compliance increases.

SECONDARY OUTCOMES:
Self-Care | The scale will be completed before the intervention and at 3, 7 and 9 weeks.
  "Chronic Dialysis Patients' Self-Care Agency (SCA)" Scores obtained from the scale are between 0-44. As the score decreases, it is evaluated as self-care power is not good.

OTHER OUTCOMES:
Patient outcomes | The Kt/V value of all patients calculated before the intervention and the change in the value measured 3, 7 and 9 weeks after the intervention will be completed by the researcher.
  "Data collection form for patients (The target Kt/V in dialysis patients is between 1.2-1.4. , Kt/V(K - urea dialyzer clearance, t - dialysis time, V - urea volume of distribution))"
Caregivers on Care Burden | The scale will be completed by the patients before the intervention and at 9th week.
  "Caregiver Burden Scale for family caregivers of hemodialysis patients" Sub-dimension scores, internal consistency of 0.87, 0.70, 0.76, 0.70, 0.70 and 0.53 indicate an increase in care burden.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Yüksel Acar, Msc, Principal Investigator — Acibadem Universty
Locations (1):
- Canan Yüksel Acar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No